CLINICAL TRIAL: NCT05956496
Title: Gingival Augmentation and Root Coverage Results With Superficial and Deep Cut Acellular Dermal Matrices
Brief Title: Gingival Augmentation and Root Coverage With Superficial and Deep Cut Acellular Dermal Matrices
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study team experienced an increased number of complications than expected
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Angela Palaiologou-Gallis, DDS, MS, Professor and Program Director, Graduate Periodontics, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC20230466H
Record Dates: First submitted 2023-07-13; First posted 2023-07-21 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Gingival Recession
Keywords: Gingival augmentation; Graft materials; Acellular dermal matrix (ADM); Subepithelial connective tissue graft (SCTG)
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Intervention Model Description: This is a split-mouth design randomized, prospective trial designed to compare two standard of care techniques.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group: Acellular Dermal Matrix - Superficial cut (ADM-S) (Placebo Comparator): A commonly used allograft material is the Acellular Dermal Matrix (ADM) which is harvested from human donor dermal tissues. Most commercially available ADM products are superficial cuts.
  Interventions: Other: Allograft Material ADM-S
- Test Group:Acellular Dermal Matrix - Deep cut (ADM-D) (Active Comparator): The use of a deep cut ADM for root coverage gingival plastic procedures.
  Interventions: Other: Allograft Material ADM-D

INTERVENTIONS:
Other: Allograft Material ADM-S — A piece of the allograft material (ADM-D) will be hydrated per the manufacturers guidelines and adapted to the recipient area after reflection of a partial thickness flap. The flap will be coronally advanced to completely cover the graft material per standard care for this procedure.
  Other Names: Acellular Dermal Matrix-superficial
  Arms: Control Group: Acellular Dermal Matrix - Superficial cut (ADM-S)
Other: Allograft Material ADM-D — A piece of the allograft material (ADM-S) will be hydrated per the manufacturers guidelines and adapted to the recipient area after reflection of a partial thickness flap. The flap will be coronally advanced to completely cover the graft material per standard care for this procedure.
  Other Names: Acellular Dermal Matrix-deep
  Arms: Test Group:Acellular Dermal Matrix - Deep cut (ADM-D)

SUMMARY:
This entire protocol involves procedures that are standard care and will randomize subjects to of one two routine care procedures. Patients needing root coverage for gingival recession will be enrolled.

DETAILED DESCRIPTION:
Each subject will be randomized to one of the treatments for the first side and the contralateral side will receive the other treatment. No risk or benefit is expected from being assigned to either group as both procedures are both standard care. In both groups, a commercially available allograft (ADM-D or ADM-S) will be used.

Allocation of subjects into test group or control group will be based on numbers drawn from a stack of sealed envelopes.

Grafting teeth with gingival recession is often done to improve esthetics and tooth sensitivity as well as prevent recession from progressing. When recession coverage procedures are done, a soft tissue graft material is inserted between the gums and the tooth to help decrease the amount of root exposure. This material is obtained from a donor and may originate from a deeper or shallower layer of the donor skin. The study team seek to determine if the origin of the graft material (deep or shallow) influences the amount of root coverage achieved.

ELIGIBILITY:
Inclusion Criteria:

* Patients between age 18 and 89
* Patients needing root coverage procedures for gingival recession in one or more teeth in the same arch bilaterally (split mouth)
* Patients must be nonsmokers, former smokers, or current smokers who smoke <10 cigarettes per day, by self-report.
* Female patients who have undergone a hysterectomy, tubal ligation, or menopause, and non- pregnant women of child-bearing potential.

Exclusion Criteria:

* Patients who disclose that they will not be able to cooperate with the follow-up schedule.
* Patients who are mentally incompetent, prisoners, or pregnant (as obtained via chart review or self-report)
* Pregnant women or women intending to become pregnant during study period.
* Smokers who smoke > 10 cigarettes per day

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2023-10-03 (Actual); Primary Completion 2024-04-09 (Actual); Study Completion 2024-04-09 (Actual)

PRIMARY OUTCOMES:
Percentage root coverage | Baseline to 12 months
  Measured as change in percentage root coverage
Keratinized tissue width | Baseline to 12 months
  Measured as change in keratinized tissue width

CONTACTS AND LOCATIONS:
Overall Officials: Angela Palaiologou-Gallis, DDS, MS, Principal Investigator — University of Texas Health Science Center San Antonio
Locations (1):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected de-identified Individual Participant data (IPD) that underlie results in a publication
Supporting Information: Study Protocol, SAP
Time Frame: When summary data are published or otherwise made available